CLINICAL TRIAL: NCT05041075
Title: Effects of Weighted Blankets on Anxiety for Pediatric Oncology Patients During Outpatient Chemotherapy Infusion
Brief Title: Effect of Weighted Blankets on Anxiety for Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-3150.cc
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WB:UC (Active Comparator): Weighted Blanket 2nd infusion Usual Care 3rd infusion
  Interventions: Device: Weighted Blanket
- UC:WB (Active Comparator): Usual Care 2nd infusion Weighted Blanket 3rd infusion
  Interventions: Device: Weighted Blanket

INTERVENTIONS:
Device: Weighted Blanket — Weighted blankets provide Deep Pressure Stimulation (DPS) or Deep Touch Pressure (DTP) which has advantages in both physical and psychological domains.

SUMMARY:
The use of weighted blankets has been studied in the adult population but there is a lack of evidence to determine their benefit among a pediatric population, specifically oncology pediatric patients. Pediatric oncology patients routinely experience anxiety during therapy and as cure rates increase, attention has progressively turned to treating psychosocial aspects of care.

DETAILED DESCRIPTION:
A randomized 2x2 cross-over design will be utilized for this study. The study team will randomize participants to one of two sequences: 1) weighted blanket first then usual care or 2) usual care first then weighted blanket. The cross-over design allows the researchers to compare both within and between group differences. The advantages of the cross-over design allow minimize potential confounding bias as patients will serve as their own controls as well as potential for adequate power with smaller patient enrollment. As this study is conducted during chemotherapy treatments, the 30-day period in between patient treatments will be considered the washout period. This timeframe between chemotherapy infusions was chosen to try to capture patients in a similar state of baseline anxiety. This helps to provide adjustments to variability but should not limit accrual based on the number of patients that get chemotherapy within a 30-day period.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed pediatric oncology patients between the ages of 4 and 17 receiving outpatient chemotherapy infusions in one of the two designated out patient locations (Anschutz Campus and Colorado Springs Hospital)
* Patients who have a "liquid tumor" (leukemia or lymphoma), "solid tumor", or a neuro-oncologic diagnosis
* Patients who can complete the CAM-S and CAM-T as proven by seriation screening.
* Patients who are great than 13.5kg in weight, due to weighted blanket size options
* Patients whose second and third outpatient chemotherapy occur within 30 days of each other.
* English and Spanish speaking

Exclusion Criteria:

* Patients who are younger than 4 years of age, or older than 17 years of age
* Relapsed patients
* Patients who are undergoing bone marrow transplant or had a previous bone marrow transplant
* Patients receiving chemotherapy infusions at North Campus and South Campus locations
* Patients in the inpatient setting
* Patients who utilize a weighted blanket at home currently or previously
* Patients who fail seriation screening during enrollment
* Patients who start initial chemotherapy infusions in the outpatient setting

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Children's Anxiety Meter-State (CAM-S) assessment | 12 months
  The CAM-S is completed by showing the child a picture of a mercury thermometer and asking the child to "Pretend that all of your worried or nervous feelings are in the very bottom down here (point to scale). If you are a little bit worried or nervous, the feelings might come up just a little bit (move finger up). If you are very, very worried, or nervous, the feelings might come up just a little bit (move finger up to the top). Put a line showing how much worry or nervousness you feel right now." This scale is from measured from 1-10. Higher values indicate higher anxiety. The CAM-S will be administered during the following times: prior to infusion start, thirty minutes into the treatment or end of the treatment if <30 minutes and end of the treatment (see Figure 1).

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory Generic Core Scales (Peds QL 4.0) | 12 months
  The Peds QL 4.0 is a 23-item questionnaire and is broken up into four sections: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). These questions are aimed to measure health-related quality of life in children and adolescents who are healthy and those with acute or chronic health conditions (Varni, Burwinkle, Seid & Skarr, 2003). We will utilize the parent-proxy questionnaires with responses measured on a 5-point response scale: 0 = never a problem; 1= almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem. The scale is recoded and summarized to have a score ranging from 0 to 100 where higher values indicate higher quality of life.

OTHER OUTCOMES:
Weighted Blanket Use | 12 months
  Prior to discharge, a trained infusion nurse or a member of the weighed blanket research team will ask participants/families to classify if the participant used the blanket 0-20%, 20-40%, 40-60%, 60-80%, or 80-100% of their total infusion time.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Olson, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No